CLINICAL TRIAL: NCT06487611
Title: The Presence of Humanoid Robot With Older Adults at Homes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Professor and Associate Head (Research), The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P0041148
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Loneliness; Cognitive Impairment; Depression; Self Efficacy; Sense of Coherence
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Intervention Model Description: This study will employ a two-arm pilot randomized control trial with qualitative interviews.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A humanoid social robot (Experimental): Project team will set up a physical robot at their homes. Each participant will be given a protocol to engage with different features of the robot every day. Participants are asked to complete the assigned daily tasks at their own homes
  Interventions: Behavioral: A humanoid social robot
- Control (No Intervention)

INTERVENTIONS:
Behavioral: A humanoid social robot — A humanoid social robot-mediated programme, including human-robot interactions, listening songs and daily news, doing physical activities and play memory games
  Arms: A humanoid social robot

SUMMARY:
Background Older adults experience significant physical, cognitive and environmental losses in their later life. Self-supported 'aging-in-place' has benefits for mental health and the quality of life for older people. In the field of gerontological nursing, person-centered holistic care highlights the importance of enabling older people and their significant others (such as older spouse or other family caregivers) to establish healthful relationships so to improve older adults' physical, psychological, mental and social wellbeing. However, globally and also most recommended by Hong Kong government, home-based care services for older adults have not been fully developed. Research on the use of robots supporting older adults is given increasing attention in the globe, but most of them were focused on aiding older adults who are living with dementia or residing in nursing homes. More robotic research needs to be conducted at their own homes in the community and support older people in having an independent lifestyle.

Study Aim This study aims to investigate the feasibility and acceptability of home-based physical robot HUMANE by community-dwelling Chinese older adults and soon-to-be-aged adults and their family caregivers.

Study design and method This study will employ a two-arm pilot randomized control trial with qualitative interviews. People aged 50 or above who are receiving home care from family members will be recruited to this study. Purposive sampling will be adopted in recruitment. The robot HUMANE will be used by the intervention group for a 6-week trial. Loneliness, cognitive function, emotional status, self-efficacy, mutuality and sense of coherence will be measured at baseline (day-1) and immediately post-intervention (week-6) to examine preliminary effect of using robot at home.

Data analysis SPSS Statistics 26 will be adopted for all analyses. Descriptive statistics, generalized estimating equations (GEE) models and a deductive content analysis approach will be used in data analysis.

Significances of the study The study will add evidences in the field that social robot may be able to address some of the unmet needs of older people living at their own homes in the community, particularly relating to loneliness, enhancing the development of home-based care services for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese aged 50 years and above;
* Need home-based care from family caregiver, including spouses;
* Live with at least one family caregiver at his/her own home (not in residential care homes) in Hong Kong;
* Are able to communicate in Cantonese.

Exclusion Criteria:

* With acute mental disorders or disabling diseases that may limit the practice of engaging with robot; and
* have limited access to electricity and this makes them hard to use technology at home.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Loneliness | at baseline (day-1) and immediately post-intervention (week-6)
  6-item Loneliness scale: It consists of two subscales: emotional loneliness (1-3 items) and social loneliness (4-6 items). There are negatively (1-3) and positively (4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. A score of 3 is the optimal cut point, with moderate or severe loneliness [score of 3-6]

SECONDARY OUTCOMES:
Memory | at baseline (day-1) and immediately post-intervention (week-6)
  5-items Abbreviated Memory Inventory for the Chinese (AMIC) scores range from 0-5 (1 point for each item; 0-best to 5-worse). An AMIC score ≥ 3 is predictive of MCI
Emotion status | at baseline (day-1) and immediately post-intervention (week-6)
  4. PHQ-2 includes 2 items. Not at all scores 0; Several days scores 1; More than half the days scores 2; and Nearly every day scores 3. Refuse to answer we put -99. A PHQ-2 score ranges from 0-6. A score of 3 is the optimal cut point, If the score is 3 or greater, major depressive disorder is likely.
Sense of coherence (SOC) | at baseline (day-1) and immediately post-intervention (week-6)
  The SOC-13 scale has three components: Comprehensibility (items 2, 6, 8, 9, 11), Manageability (items 3, 5, 10, 13) and Meaningfulness (items 1, 4, 7, 12). This scale is rated on a 7-point likert scale, a total score can also be used and the coding for items 1, 2, 3, 7 and 10 should be reversed. SOC scores range from 13 to 91
Self-efficacy | at baseline (day-1) and immediately post-intervention (week-6)
  The Chinese version of the General Self-Efficacy Scale is a reliable and valid scale that can be used with confidence in community Chinese soon-to-be-aged adults. The Scale consists of 10 items that measure a generalized sense of competence. All items are rated on a 4-point Likert scale ranging from 1='Not at all true' to 4='Exactly true'. The higher the score, the greater self-efficacy the respondents possess.
mutuality (if applicable) | at baseline (day-1) and immediately post-intervention (week-6)
  Each item is scored on a 5-point Likert-type scale from 0 ( not at all ) to 4 ( a great deal ). The total scale score, a mean of all item scores, ranges from 0 to 4: higher scores means greater mutuality.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will only be available per request and approve by the study team. The study team will publish the research findings without individual recognized data

REFERENCES:
- [Derived] Zhao IY, Leung AYM, Huang Y, Liu Y. A Social Robot in Home Care: Acceptability and Utility Among Community-Dwelling Older Adults. Innov Aging. 2025 Mar 8;9(5):igaf019. doi: 10.1093/geroni/igaf019. eCollection 2025. PMID 40386025

DOCUMENTS (1):
  • Study Protocol (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT06487611/Prot_000.pdf